CLINICAL TRIAL: NCT02854839
Title: Multi-center, Open, Phase 2a Clinical Trial to Evaluate the Efficacy and Safety of MG4101 in Hepatocellular Carcinoma After TACE
Brief Title: A Study of MG4101 (Allogeneic Natural Killer Cell) for Intermediate-stage of Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MG4101-HCC-P2a
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2018-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Control Group (No Intervention): Patients will be randomized 1:1 to the control group and the treatment group. Patients who had allocated control group will not receive adjuvant treatment.
- The Treatment Group (MG4101) (Experimental): Patients will be randomized 1:1 to the control group and the treatment group. The treatment group will receive 6 times of MG4101(allogeneic natural killer cells) on week 0, 1, 2, 5, 6, 7.
  Interventions: Biological: MG4101

INTERVENTIONS:
Biological: MG4101 — MG4101 is ex vivo-expanded, allogeneic natural killer cells. MG4101 were manufactured from normal healthy donor who underwent lymphopheresis under good manufacturing practice (GMP) conditions.
  Other Names: allogeneic natural killer cells
  Arms: The Treatment Group (MG4101)

SUMMARY:
The propose of this study is evaluate the safety and efficacy of MG4101 (allogeneic Natural killer cells) in patients with hepatocellular carcinoma (HCC) after transarterial chemoembolization (TACE).

DETAILED DESCRIPTION:
This is randomized, multi-center, open-labeled, Phase 2a study in patients with HCC after transarterial chemoembolization (TACE). A total of 78 patients will be randomized(1:1) into one of the two group, to receive adjuvant therapy using MG4101 (allogeneic Natural killer cells, Treatment group) or no adjuvant therapy (Control group).

Patients who were assigned Treatment group will receive 2 cycles of MG4101 (each cycle is 3 treatments at a frequency of once per week, between each cycle has 3 weeks of withdrawal period). After treatment period, patients will undergo follow up for progression and survival every 12 weeks (± 7 days) and follow up 1 year after the last patient's enrollment date.

The Control group's patients will will undergo follow up for progression and survival every 12 weeks (± 7 days) and follow up 1 year after the last patient's enrollment date.

ELIGIBILITY:
Inclusion criteria

1. Patients who are between 20 to 80 years of age
2. Life expectancy > 12 weeks
3. Patients have complete remission according to the mRECIST by Dynamic contrast-enhanced 3- or 4-phase CT or tissue biopsy

   * Patients were diagnosed Hepatocellular Carcinoma BCLC stage B be-fore TACE.
   * Dynamic contrast-enhanced CT must be within 4 weeks after the TACE.
4. Previous TACE with the following:

   * Lipiodol mixed with chemotherapy (such as adriamycin etc.)
   * Used with Gelatin sponge or Polyvinyl alcohol or microsphere.
5. Patients who had local treatment such as Resection, Radiofrequency Ablation, Percutaneous ethanol injection and Transarterial chemoembolization can participates study.
6. Patients whose Child-Pugh score is less than B8.
7. Patients whose ECOG score is 0
8. Patients who satisfy the following conditions of the blood test, kidney function test, and liver function test.

   * Absolute neutrophil count ≥ 1,000 x 10^6 /L
   * hemoglobin level ≥ 8.5 g/㎗
   * platelet count ≥ 50,000 /㎣
   * Total bilirubin < 3.0 ㎎/㎗
   * Serum creatinine ≤ 1.5 x upper normal limit (UNL)
   * Total Albumin ≥ 2.8 ㎎/㎗
9. Able and willing to provide written informed consent and to comply with the study protocol.

Exclusion criteria

1. Patients who have metastasis.
2. Patients who have Portal vein or hepatic vein invasion.
3. Patient with medical history for the following:

   * Patients with Living donor Liver Transplantation or Orthotopic liver transplantation.
   * Patients who have received anti-cancer chemotherapy for 4 weeks prior to the study.
   * Patients who have not recovered adverse reaction prior to the study.
   * Patients who have received external beam radiation on liver, immunotherapy, cell therapy, and target therapy.
   * Prior use of systemic anticancer chemotherapy twice.
4. Patients who have a history of malignant tumors in 5 years prior to the study with the exception of Carcinoma in situ..
5. Patients who have a history of autoimmune disease such as Rheuma-toid arthritis, systemic Lupus Erythematosus, Vasculitis, Multiple sclerosis, Adolescent Insulin-dependent Diabetes Mellitus, etc.
6. Patients who have history of human immunodeficiency virus (HIV) infection.
7. Patients who have participated in other clinical trials within 4 weeks prior to this study.
8. Patients who treated with immunosuppressant for 3 months prior to this study.
9. Patients who have any condition that was uncontrolled or needed treatment.
10. Pregnant or breast-feeding subjects.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Time To progression | every 12 weeks, up to the time of death or 18 months

SECONDARY OUTCOMES:
Progression-free survival | every 12 weeks, up to the time of death or tumor progression, up to 18 months
Overall survival | every 12 weeks, up to the time of death, up to 18 months
change of Tumor Markers(AFP, Alpha-Fetoprotein) | every 12 weeks, up to the time of death or tumor progression, up to 18 months
Safety of MG4101 as evaluated by Incidence of adverse events (AEs), serious adverse events (SAEs) | up tp 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hwan Yoon, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - Seoul National University Hospital, Seoul
  - Seoul Asan Medical center, Seoul
  - Samsung Medical Center, Seoul
  - Korea Univ. Guro Hospital, Seoul
  - Severance hospital, Seoul
  - Ajou Univ. Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Undecided